CLINICAL TRIAL: NCT02232178
Title: A Randomized, Blinded, Inpatient Study to Investigate the PK, Relative Bioavailability and Safety of 2 Doses of XaraColl (200 and 300 mg Bupivacaine HCl) Compared to Bupivacaine HCl Infiltration (150 mg) After Open Laparotomy Hernioplasty
Brief Title: Pharmacokinetics, Relative Bioavailability and Safety of Xaracoll Implant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: INN-CB-013
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Hernioplasty
Keywords: unilateral inguinal hernioplasty
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 100mg Xaracoll implants (Experimental): Bupivacaine HCl implant
  Interventions: Drug: 2 100mg Xaracoll implants
- 3 100mg Xaracoll implants (Experimental): Bupivacaine HCl implant
  Interventions: Drug: 3 100mg Xaracoll implants
- 150mg Bupivacaine HCl injection (Active Comparator): Bupivacaine HCl
  Interventions: Drug: 150mg Bupivacaine HCl injection

INTERVENTIONS:
Drug: 2 100mg Xaracoll implants
  Other Names: Bupivacaine HCl implant
  Arms: 2 100mg Xaracoll implants
Drug: 3 100mg Xaracoll implants
  Other Names: Bupivacaine HCl implant
  Arms: 3 100mg Xaracoll implants
Drug: 150mg Bupivacaine HCl injection
  Other Names: Bupivacaine HCl
  Arms: 150mg Bupivacaine HCl injection

SUMMARY:
Assess the pharmacokinetic profile of 2 doses of the XaraColl® implant after open laparotomy hernioplasty and assess the relative bioavailability of Xaracoll compared to a local bupivacaine infiltration.

DETAILED DESCRIPTION:
Inguinal hernioplasty is a common surgery. Common surgical methods used include laparoscopic and open placement of synthetic mesh. Managing postoperative pain and preventing morbidity after open mesh hernioplasty remain considerable medical challenges.

Bupivacaine is a local anesthetic (pain medicine) that has an established safety profile. Collagen is a protein that is found in all mammals. The Xaracoll implant is a thin flat sponge made out of collagen that comes from cow tendons and contains bupivacaine. When inserted into a surgical site, the collagen breaks down and bupivacaine is released at the surgical site to provide postoperative pain control.

This study will assess the pharmacokinetic profile of 2 doses of the XaraColl implant after open laparotomy hernioplasty and assess the relative bioavailability of the Xaracoll implant compared to a local bupivacaine infiltration.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman who is ≥ 18 years of age
2. Has a planned unilateral inguinal hernioplasty (open laparotomy, tension free technique)
3. If female, is nonpregnant

Exclusion Criteria:

1. Scheduled for bilateral inguinal hernioplasty or other significant concomitant surgical procedures
2. Has undergone major surgery within 3 months of the scheduled hernioplasty or plans to undergo another laparotomy procedure within 30 days postoperatively
3. Has any clinically significant unstable cardiac, neurological, immunological, renal, hepatic or hematological disease or any other condition that, in the opinion of the investigator, could compromise the patient's welfare, ability to communicate with the study staff or otherwise contraindicate study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Niebler, D.O., Study Director — Innocoll
Locations (5):
- United States (5):
  - Pinnacle Research Group, Anniston, Alabama
  - Shoals Medical Trials, Sheffield, Alabama
  - Wexner Medical Center at Ohio State University, Columbus, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - Victory Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 100mg Xaracoll Implants: Bupivacaine HCl implant
  2 100mg Xaracoll implants
- 3 100mg Xaracoll Implants: Bupivacaine HCl implant
  3 100mg Xaracoll implants
- 150mg Bupivacaine HCl Injection: Bupivacaine HCl
  150mg Bupivacaine HCl injection
Period: Overall Study
Arm/Group | 2 100mg Xaracoll Implants | 3 100mg Xaracoll Implants | 150mg Bupivacaine HCl Injection
Started | 26 | 25 | 13
Per Protocol PK Population | 26 | 24 | 11
Safety Population | 26 | 24 | 12
Completed | 25 | 24 | 12
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — ineligibility | 0 | 0 | 1
Not completed — surgical complication | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: all randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 100mg Xaracoll Implants | 3 100mg Xaracoll Implants | 150mg Bupivacaine HCl Injection | Total
Number analyzed (Participants) | 26 | 25 | 13 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.93) | 46.1 (11.40) | 48.2 (12.76) | 45.2 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 24 | 25 | 12 | 61
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 13 | 64

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum drug plasma concentration
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 72, and 96 hours after surgery.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 2 100mg Xaracoll Implants | 3 100mg Xaracoll Implants | 150mg Bupivacaine HCl Injection
Number analyzed (Participants) | 26 | 24 | 11
ng/mL | 340.4 (111.05) | 524.8 (146.45) | 348.4 (184.02)

2. Primary Outcome: AUC0-last
Description: Area under the plasma concentration-time curve from Time 0 to time of last quantifiable plasma concentration.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 72, and 96 hours after surgery.
Measure: Mean (Standard Deviation); unit: ng/mL∙hr
Arm/Group | 2 100mg Xaracoll Implants | 3 100mg Xaracoll Implants | 150mg Bupivacaine HCl Injection
Number analyzed (Participants) | 26 | 24 | 11
ng/mL∙hr | 10793.449 (5523.4326) | 18589.907 (7841.1973) | 8323.188 (4312.1940)

3. Primary Outcome: Tmax
Description: Time to maximum plasma concentration.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 72, and 96 hours after surgery.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2 100mg Xaracoll Implants | 3 100mg Xaracoll Implants | 150mg Bupivacaine HCl Injection
Number analyzed (Participants) | 26 | 24 | 11
hours | 7.271 (10.8603) | 8.567 (10.2484) | 8.783 (01.8761)

4. Primary Outcome: t1/2 (Hour)
Description: Terminal half-life.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, 48, 72, and 96 hours after surgery.
Population: Per protocol PK population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2 100mg Xaracoll Implants | 3 100mg Xaracoll Implants | 150mg Bupivacaine HCl Injection
Number analyzed (Participants) | 26 | 24 | 11
hours | 16.922 (7.6260) | 18.058 (7.6699) | 8.819 (4.5292)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 2 100mg Xaracoll Implants | 3 100mg Xaracoll Implants | 150mg Bupivacaine HCl Injection
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 21/26 | 15/24 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 100mg Xaracoll Implants (N=26) | 3 100mg Xaracoll Implants (N=24) | 150mg Bupivacaine HCl Injection (N=12)
constipation (Gastrointestinal disorders) | 6 (6) | 3 (3) | 2 (2)
nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
post procedural oedema (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1)
procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
somnolence (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1)
penile haemorrhage (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
testicular pain (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
abdominal distention (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
catheter site pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
wound infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) — Separation of the edges of the wound. There was no evidence of loss of fascial integrity.
wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
testicular oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
incisional drainage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
post procedural drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
results of the multicenter study had to be published prior to the publication of any site specific data.